CLINICAL TRIAL: NCT04254653
Title: Test of a Culturally Tailored Diabetes Nutrition Education Program for Tribal and Urban American Indian and Alaska Native (AIAN) Communities
Brief Title: Diabetes Nutrition Education for American Indian and Alaska Native Communities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-2269
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): Participants receive diabetes nutrition education classes immediately.
  Interventions: Behavioral: American Indian and Alaska Native What Can I Eat?
- Wait list intervention (Experimental): Participants wait listed (control) for 3 months and then receive the diabetes nutrition education classes.
  Interventions: Behavioral: American Indian and Alaska Native What Can I Eat?

INTERVENTIONS:
Behavioral: American Indian and Alaska Native What Can I Eat? — Participants will engage in 5 ~90 minute diabetes nutrition education classes. They will learn about healthy eating for type 2 diabetes management. Classes include didactic lesson, hands on learning activity, sharing session, mindful nutrition practice, and physical activity

SUMMARY:
This study involves pilot testing a newly developed diabetes nutrition education program for American Indian and Alaska Native adults with T2D. The first phase of this study (COMIRB Protocol 18-006) included a qualitative needs assessment to inform the development of this program. The Study Aims include: piloting the newly adapted program at 6 AI/AN collaborating sites to gain feedback on satisfaction, likability, usability and clinical outcomes such as HgA1C (measure of blood sugar control), blood pressure, and body mass index (BMI).

DETAILED DESCRIPTION:
This study involves pilot testing a newly developed diabetes nutrition education program for American Indian and Alaska Native adults with T2D. The first phase of this study (COMIRB Protocol 18-006) included a qualitative needs assessment to inform the development of this program. The second phase involves pilot testing the study at 6 collaborating AI/AN sites across the US. The Study Aims include: piloting the newly adapted program at 6 AI/AN collaborating sites to gain feedback on satisfaction, likability, usability and clinical outcomes such as HgA1C (measure of blood sugar control), blood pressure, and body mass index (BMI).

ELIGIBILITY:
Inclusion Criteria:

* AI/AN status (self-reported)
* age > 18 years
* fluent in English
* a current diagnosis of T2DM.

Exclusion Criteria:

* a major medical issue that may interfere with participation (e.g., prior cardio- or cerebrovascular disease including a recent myocardial infarction or major stroke; cancer not in remission; dialysis; active alcohol and/or substance abuse.)
* a planned move from the area within the 3 to 6 month data collection time period that would not allow completion of all the study visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate diabetes nutrition education program impact on HgA1C | 3 months for immediate intervention group 6 months for wait list control group
  Participants will have 2 A1C checks for Immediate intervention and 3 for wait list control. Immediate will have A1C tested at baseline and after the 5th class (at 3 months from baseline). Wait list will have A1C checked baseline, immediately before class #1 (3 months after baseline) and after class #5 (6 months after baseline). A1C will be checked per standard of care at the clinical site
Evaluate diabetes nutrition education program impact on blood pressure | 3 months for immediate intervention group 6 months for wait list control group
  Participants will have 3 BP checks for Immediate intervention and 5 for wait list control. Immediate will have BP tested at baseline, after the 4th class, and after the 5th class (at 3 months from baseline). Wait list will have BP checked baseline, immediately before class #1 (3 months after baseline), 1 month after baseline, after class #4, and after class #5 (6 months after baseline). Blood pressure will be checked per standard of care at the clinical site.
Evaluate diabetes nutrition education program impact on weight | 3 months for immediate intervention group 6 months for wait list control group
  Participants will have 3 weight checks for Immediate intervention and 5 for wait list control. Immediate will have weight tested at baseline, after the 4th class, and after the 5th class (at 3 months from baseline). Wait list will have weight checked baseline, at one month of wait list, immediately before class #1 (3 months after baseline), after class #4, and after class #5 (6 months after baseline). Weight will be checked per standard of care at the clinical site.
Evaluate diabetes nutrition education program impact on eating behavior | 3 months for immediate intervention group 6 months for wait list control group
  Participants will take a self-reported survey measuring their dietary habits using a food frequency table at several timepoints. Immediate intervention participants will take the survey 3 times (baseline, after class 4, after class 5). Wait list control participants will take the survey 5 times (baseline, at 1 month after baseline wait list, immediately before class #1, after class #4, after class #5)
Evaluate diabetes nutrition education program impact on nutrition knowledge | 3 months for immediate intervention group 6 months for wait list control group
  Participants will take a self-reported survey measuring their nutrition knowledge using a food frequency table at several timepoints. Immediate intervention participants will take the survey 3 times (baseline, after class 4, after class 5). Wait list control participants will take the survey 5 times (baseline, at 1 month after baseline wait list, immediately before class #1, after class #4, after class #5)
Evaluate diabetes nutrition education program impact on self efficacy for healthful eating | 3 months for immediate intervention group 6 months for wait list control group
  Participants will take a self-reported survey measuring their self efficacy for healthy eating using a food frequency table at several timepoints. Immediate intervention participants will take the survey 3 times (baseline, after class 4, after class 5). Wait list control participants will take the survey 5 times (baseline, at 1 month after baseline wait list, immediately before class #1, after class #4, after class #5)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly R Moore, MD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - Lakeport Tribal Health Consortium, Lakeport, California
  - Cherokee Indian Hospital, Cherokee, North Carolina
  - Indian Health Care Resource Center of Tulsa, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: No